CLINICAL TRIAL: NCT00720915
Title: A Cohort Study to Test That There is a Low Risk of Recurrent VTE in Patients With a First Episode of Unprovoked VTE Who Stop Anticoagulant Therapy After 3 Months of Treatment in Response to Negative D-dimer Testing
Brief Title: D-dimer to Select Patients With First Unprovoked Venous Thromboembolism Who Can Have Anticoagulants Stopped at 3 Months
Acronym: DODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMG-2007-DODS
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: unprovoked deep vein thrombosis; unprovoked pulmonary embolism; anticoagulant therapy
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Anticoagulant Therapy (Other): No Anticoagulant Therapy
  Interventions: Other: Discontinue anticoagulant therapy (Negative d-dimer)
- Anticoagulant Therapy (Other): Continue on anticoagulant therapy
  Interventions: Other: Continue on anticoagulant therapy (positive d-dimer)

INTERVENTIONS:
Other: Discontinue anticoagulant therapy (Negative d-dimer) — Patients with negative d-dimer discontinue long-term anticoagulant therapy.
  Arms: No Anticoagulant Therapy
Other: Continue on anticoagulant therapy (positive d-dimer) — Patients with positive d-dimer continue or re-start on anticoagulant therapy
  Arms: Anticoagulant Therapy

SUMMARY:
The purpose of this study is to determine if the risk of recurrent venous thromboembolism (VTE) after stopping therapy is low and acceptable in patients with a first unprovoked proximal deep vein thrombosis (DVT) or pulmonary embolism (PE) who have completed 3 months of therapy and who have a negative D-dimer test on therapy and 1 month after stopping therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be >= 18 years of age
2. Have had ONE episode of unprovoked proximal DVT and/or PE
3. Have completed 3 uninterrupted months of warfarin therapy (target INR of 2.0-3.0)

Exclusion Criteria:

1. Another indication for long-term anticoagulation (e.g., atrial fibrillation)
2. A high risk of bleeding as evidenced by any of the following:

   * Age greater than 75 years
   * Previous episode of major bleeding where the cause was not effectively treated
   * Known chronic thrombocytopenia with a platelet count of less than 120,000 x 10^9 /L
   * Known chronic renal impairment with a creatinine of more than 150 mumols /litre (1.7 mg/dl)
   * Known chronic liver disease with a total bilirubin of more than 25 mumols /litre (1.5 mg/dl)
   * Active peptic ulcer disease
   * Poor compliance with, or control of, anticoagulant therapy during initial treatment
   * Requires dual antiplatelet therapy (e.g. aspirin and clopidogrel)
3. A vena caval filter
4. Has had D-dimer testing performed within 2 months of potential enrollment other than for evaluation of suspected recurrent VTE that was not confirmed
5. Has a life expectancy less than 5 years
6. Is unable to attend follow-up visits because of geographic inaccessibility
7. Is participating in a competing clinical investigation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2008-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Suspected Recurrent DVT | up to 7 years
Suspected (recurrent) pulmonary embolism | up to 7 years
Bleeding | up to 7 years
Death | up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MB MRCP(I) FRCP(C) PhD, Principal Investigator — McMaster University
Locations (13):
- United States (7):
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Centre, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - UNC Thrombophilia Program, Chapel Hill, North Carolina
  - Intermountain Medical Centre, Murray, Utah
- Canada (4):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - St. Joseph's Health Care Centre, Hamilton, Ontario
  - Henderson Hospital, Hamilton, Ontario
- Limerick, Mid Western Regional Hospital, Limerick, Ireland
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Kearon C, Parpia S, Spencer FA, Schulman S, Stevens SM, Shah V, Bauer KA, Douketis JD, Lentz SR, Kessler CM, Connors JM, Ginsberg JS, Spadafora L, Julian JA. Long-term risk of recurrence in patients with a first unprovoked venous thromboembolism managed according to d-dimer results; A cohort study. J Thromb Haemost. 2019 Jul;17(7):1144-1152. doi: 10.1111/jth.14458. Epub 2019 May 20. PMID 31033194
- [Derived] Kearon C, Parpia S, Spencer FA, Baglin T, Stevens SM, Bauer KA, Lentz SR, Kessler CM, Douketis JD, Moll S, Kaatz S, Schulman S, Connors JM, Ginsberg JS, Spadafora L, Bhagirath V, Liaw PC, Weitz JI, Julian JA. Antiphospholipid antibodies and recurrent thrombosis after a first unprovoked venous thromboembolism. Blood. 2018 May 10;131(19):2151-2160. doi: 10.1182/blood-2017-09-805689. Epub 2018 Feb 28. PMID 29490924
- [Derived] Kearon C, Spencer FA, O'Keeffe D, Parpia S, Schulman S, Baglin T, Stevens SM, Kaatz S, Bauer KA, Douketis JD, Lentz SR, Kessler CM, Moll S, Connors JM, Ginsberg JS, Spadafora L, Julian JA; D-dimer Optimal Duration Study Investigators. D-dimer testing to select patients with a first unprovoked venous thromboembolism who can stop anticoagulant therapy: a cohort study. Ann Intern Med. 2015 Jan 6;162(1):27-34. doi: 10.7326/M14-1275. PMID 25560712